CLINICAL TRIAL: NCT07295002
Title: COmpletion Sentinel Node Resection With or Without Minimally invAsive and Endoscopic Cooperative Surgery Following noncuRative Endoscopic Submucosal Dissection for Early Gastric Cancer
Brief Title: Sentinel Node Resection With or Without LECS After Noncurative ESD for EGC
Acronym: Co-SNARE
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Region Stockholm (Other Government)
Responsible Party: Principal Investigator, Ioannis Rouvelas, Principal Investigator, MD, PhD, Region Stockholm
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2025-05956-01
Record Dates: First submitted 2025-11-15; First posted 2025-12-19 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Early Gastric Cancer
Keywords: sentinel node-resection; minimal invasive surgery
MeSH Terms: conditions — Stomach Neoplasms | interventions — Laparoscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ICG-guided lymphadenectomy +/- LECS (Experimental): Laparoscopic and endoscopic cooperative surgery to locally resect the gastric scar. This method will we be used for cases where pathology showed positive vertical margin after ESD. Otherwise, submucosal injection of ICG in quadrants around the scar after ESD, followed by laparoscopic resection of positive lymph nodes after 15 minutes
  Interventions: Procedure: ICG-guided lymphadenectomy; Procedure: Laparoscopic and endoscopic cooperative surgery (LECS)

INTERVENTIONS:
Procedure: ICG-guided lymphadenectomy — Submucosal injection of ICG in quadrants around the scar after ESD, followed by laparoscopic resection of positive lymph nodes after 15 minutes
Procedure: Laparoscopic and endoscopic cooperative surgery (LECS) — Endoscopic marking and submucosal cutting around the scar after ESD, followed by perforation of the gastric wall and laparoscopic full thickness resection of the area under endoscopic guidance.

SUMMARY:
For patients with non-curative resection after endoscopic submucosal dissection (ESD) for early gastric cancer (EGC), complementary surgery is generally recommended. However, about 2/3 of patients have no remaining tumor in the stomach or regional lymph nodes. In this trial, Indocyanine Green (ICG)-guided lymphadenectomy with or without laparoscopic and endoscopic cooperative surgery (LECS) will be tested as a less invasive alternative in such cases. For patients with a primary radically resected EGC, ICG-guided lymphadenectomy alone will be performed. For patients with deep-margin positive EGC, ICG-guided lymphadenectomy and LECS will be performed, in order to ensure both local tumor control in the stomach and in regional nodes.

DETAILED DESCRIPTION:
Endoscopic submucosal dissection (ESD) is the recommended treatment for early gastric cancer (EGC) who are fullfillling the criteria based on international guidelines. After ESD, some resections are classified as non-curative because of factors such as non radicality (especially when the deep margin is positive for cancer), lymphovascular invasion or deep submucosal invasion Sm>1. In such cases, guidelines recommend complementary gastrectomy and lymphadenectomy. Gastrectomy is known to carry a risk for severe complications in about 9-22 % of cases. Furthermore, up to 2/3 of patients are found to have no remaining tumor in the stomach or regional nodes after surgery.

In this trial, Indocyanine Green (ICG)-guided lymphadenectomy including sentinel node resection, with or without complementary laparoscopic and endoscopic cooperative surgery (LECS) will be tested as a less invasive treatment option. For patients with radically resected EGC, ICG-guided lymphadenectomy alone will be performed. In patients with deep margin positive EGC, ICG-guided lymphadenectomy and LECS will be performed.

ICG-guided lymphadenectomy is performed by first injecting 100 times diluted ICG in four quadrants in the submucosa around the tumor scar with gastroscopy. After 15 minutes, the draining nodes will be visualized with laparoscopy, and locally resected. LECS is performed by endoscopic marking of the scar followed circumferential mucosal cutting, trimming, and perforation of the stomach followed by full-thickness resection of the scar with laparoscopy. After resection, the resected specimen will be taken out and the stomach defect sutured laparoscopically.

After the procedure, the patient will be presented at a multidisciplinary tumor board. If only clinical follow-up is recommended, the patient will be followed closely with gastroscopy and computer tomography (CT) scan every 3 months for the first year.

ELIGIBILITY:
Inclusion Criteria:

* EGC previously treated with ESD according to current guidelines (differentiated adenocarcinoma, not ulcerative, of any size, differentiated adenocarcinoma ulcerative </=3cm, undifferentiated adenocarcinoma not ulcerative </=2cm)
* Non curative resection

  * Lymphovascular invasion
  * Non-radical resection vertical margin
  * deep submucosal invasion
* Signed informed consent

Exclusion Criteria:

* Location within 2 cm from cardia or pylorus
* Non-curative resection with only non-radicality horizontal margin
* Inoperative because of severe comorbidities
* Previous radiotherapy to the upper abdomen
* Pregnancy
* Allergy to ICG
* Inability to provide informed consent due to cognitive impairment, language barrier, or other reasons impairing understanding and autonomous decision-making.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2029-10-01 (Estimated); Study Completion 2029-10-01 (Estimated)

PRIMARY OUTCOMES:
Severe complications defined as Clavien-Dindo >/= III | Periprocedural
  Safety of the procedure, defined as Clavien-Dindo complication grade >/= III

SECONDARY OUTCOMES:
Any complications | Periprocedural
  Any complication during the procedure (Clavien-Dindo II-IV)
Postoperative bleeding | Periprocedural
  Postoperative bleeding requiring blood transfusion
Leakage | Periprocedural
  Leakage/postoperative abscess requiring drainage
Operation time | Periprocedural
  Time of the surgical procedure
Pathological tumor (T)-stage | Up to 2 months post procedure
  Depth of tumor invasion into the gastric wall (for LECS cases)
Tumor-free resection margins | Up to 2 months post procedure
  The rate of horizontal and vertical margins free of tumor cells (for LECS cases).
Number of lymph nodes | Periprocedural
  Number of lymph nodes harvested during the procedure
Number of positive lymph nodes | Up to 2 months post procedure
  Number of lymph nodes positive for cancer
Hospital-stay | From the day of the procedure until patient is discharged from the hospital, assessed up to 12 weeks post procedure
  Number of days from the procedure until discharge
Health-related quality of life (HQL) score QLQ-30 | Preoperatively, after 30 days and 1 year
  Pre and postoperative HQL, tested with the validated score QLQ-C30 (The EORTC QLG Core Questionnaire for cancer patients)
Health-related quality of life (HQL) score OG25 | Preoperatively, after 30 days and 1 year
  Pre and postoperative HQL, tested with the validated score OG25 (The EORTC QLG Module Questionnaire specifically for esophago-gastric patients)
30-day mortality | From procedure to maximum 30 days postoperatively
  30-day mortality
In-hospital mortality | From the day of the procedure until patient is discharged from the hospital, assessed up to 12 weeks post procedure
  In-hospital mortality
1-year disease-free survival | Until 1 year after the procedure
  1-year disease-free survival

CONTACTS AND LOCATIONS:
Overall Officials: Ioannis Rouvelas, MD, PhD, Principal Investigator — ME Övre buk, Karolinska Universitetssjukhuset
Locations (1):
- Karolinska University Hospital Huddinge, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Belia F, Biondi A, Agnes A, Santocchi P, Laurino A, Lorenzon L, Pezzuto R, Tirelli F, Ferri L, D'Ugo D, Persiani R. The Use of Indocyanine Green (ICG) and Near-Infrared (NIR) Fluorescence-Guided Imaging in Gastric Cancer Surgery: A Narrative Review. Front Surg. 2022 Jun 28;9:880773. doi: 10.3389/fsurg.2022.880773. eCollection 2022. PMID 35836598
- [Background] Morais R, Libanio D, Dinis Ribeiro M, Ferreira A, Barreiro P, Bourke MJ, Gupta S, Amaro P, Kuttner Magalhaes R, Cecinato P, Boal Carvalho P, Pinho R, Rodriguez de Santiago E, Sferrazza S, Lemmers A, Figueiredo M, Pioche M, Gallego F, Albeniz E, Ramos Zabala F, Uchima H, Berr F, Wagner A, Marques M, Pimentel-Nunes P, Goncalves M, Mascarenhas A, Soares EG, Xavier S, Faria-Ramos I, Sousa-Pinto B, Gullo I, Carneiro F, Macedo G, Santos-Antunes J. Predicting residual neoplasia after a non-curative gastric ESD: validation and modification of the eCura system in the Western setting: the W-eCura score. Gut. 2023 Dec 7;73(1):105-117. doi: 10.1136/gutjnl-2023-330804. PMID 37666656
- [Background] van den Boorn HG, Stroes CI, Zwinderman AH, Eshuis WJ, Hulshof MCCM, van Etten-Jamaludin FS, Sprangers MAG, van Laarhoven HWM. Health-related quality of life in curatively-treated patients with esophageal or gastric cancer: A systematic review and meta-analysis. Crit Rev Oncol Hematol. 2020 Oct;154:103069. doi: 10.1016/j.critrevonc.2020.103069. Epub 2020 Aug 5. PMID 32818901
- [Background] Tsekrekos A, Vossen LE, Lundell L, Jeremiasen M, Johnsson E, Hedberg J, Edholm D, Klevebro F, Nilsson M, Rouvelas I. Improved survival after laparoscopic compared to open gastrectomy for advanced gastric cancer: a Swedish population-based cohort study. Gastric Cancer. 2023 May;26(3):467-477. doi: 10.1007/s10120-023-01371-8. Epub 2023 Feb 19. PMID 36808262
- [Background] Nevo Y, Goldes Y, Barda L, Nadler R, Gutman M, Nevler A. Risk Factors for Complications of Total/Subtotal Gastrectomy for Gastric Cancer: Prospectively Collected, Based on the Clavien-Dindo Classification System. Isr Med Assoc J. 2018 May;20(5):277-280. PMID 29761671
- [Background] Wang WJ, Li HT, Yu JP, Su L, Guo CA, Chen P, Yan L, Li K, Ma YW, Wang L, Hu W, Li YM, Liu HB. Severity and incidence of complications assessed by the Clavien-Dindo classification following robotic and laparoscopic gastrectomy for advanced gastric cancer: a retrospective and propensity score-matched study. Surg Endosc. 2019 Oct;33(10):3341-3354. doi: 10.1007/s00464-018-06624-7. Epub 2018 Dec 17. PMID 30560498
- [Background] Japanese Gastric Cancer Association. Japanese Gastric Cancer Treatment Guidelines 2021 (6th edition). Gastric Cancer. 2023 Jan;26(1):1-25. doi: 10.1007/s10120-022-01331-8. Epub 2022 Nov 7. PMID 36342574
- [Background] Pimentel-Nunes P, Libanio D, Bastiaansen BAJ, Bhandari P, Bisschops R, Bourke MJ, Esposito G, Lemmers A, Maselli R, Messmann H, Pech O, Pioche M, Vieth M, Weusten BLAM, van Hooft JE, Deprez PH, Dinis-Ribeiro M. Endoscopic submucosal dissection for superficial gastrointestinal lesions: European Society of Gastrointestinal Endoscopy (ESGE) Guideline - Update 2022. Endoscopy. 2022 Jun;54(6):591-622. doi: 10.1055/a-1811-7025. Epub 2022 May 6. PMID 35523224
- [Background] Murakami T. Early cancer of the stomach. World J Surg. 1979 Nov;3(6):685-92. doi: 10.1007/BF01654788. No abstract available. PMID 532187

DOCUMENTS (1):
  • Study Protocol (2025-09-02): https://cdn.clinicaltrials.gov/large-docs/02/NCT07295002/Prot_000.pdf